CLINICAL TRIAL: NCT03052920
Title: Cochlear Implantation in Adults With Asymmetric Hearing Loss Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Midwest Ear Institute (Other); House Clinic, Inc. (Industry); NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201612147
Record Dates: First submitted 2017-02-09; First posted 2017-02-14 (Actual); Results first posted 2021-10-18 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Hearing Loss
Keywords: cochlear implant; asymmetric hearing loss
MeSH Terms: conditions — Hearing Loss | interventions — Cochlear Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Cochlear Implantation (Experimental): Cochlear implantation of the poor hearing ear
  Interventions: Device: Cochlear implant

INTERVENTIONS:
Device: Cochlear implant — Participants who have failed a BiCROS or bilateral hearing aid trial and otherwise meet inclusion criteria will receive a cochlear implant at the poor hearing ear. Post-implant, participants will continue use of a hearing aid at the better ear and the cochlear implant at the poor ear.
  Other Names: Cochlear America; Advanced Bionics; MED-EL

SUMMARY:
This longitudinal study evaluates the possible benefit of cochlear implantation in the poor ear of adults with asymmetric hearing loss who continue to use a hearing aid in the better hearing ear.

DETAILED DESCRIPTION:
The study will be conducted as a multicenter, prospective, single-arm clinical trial, evaluating the efficacy and safety of cochlear implantation in patients with asymmetric hearing loss. A repeated-measures analysis will be employed whereby patients will act as their own controls. Participants will be recruited from surgeons and audiologists in Otolaryngology departments at the participating sites.

Participants will be evaluated at multiple intervals using a variety of test measures (addressing sound localization, understanding speech in noise, understanding speech in quiet, and quality of life).

Prior to receiving a cochlear implant (CI) in the poor hearing ear, participants will be evaluated as follows:

* Hearing aid (HA) in the better ear alone
* HA in the poor ear alone
* Bilateral HAs

Participants who have not previously used a poor-ear hearing aid or BiCROS hearing aid will complete a 1-2 week trial and be evaluated at the end of the trial. If performance is better with the alternate therapy (bilateral hearing aids or BiCROS hearing aid) than the better ear alone performance and the participant prefers the alternate therapy, the participant will not continue in the study.

Participants who do continue in the study will be evaluated at several post-implant intervals. Post-implant evaluations will occur at 3, 6, 9, and 12 months after initial stimulation of the CI. Participants will be evaluated as follows:

* HA in the better ear alone
* CI in the poor ear alone
* HA and CI together

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* English as the native language
* Have a desire for functional binaural hearing
* Have failed a previous hearing aid (HA) treatment for asymmetric hearing loss (BiCROS or poor ear HA) or willing to complete a trial if necessary
* Willingness to comply with all study requirements
* Ability to provide informed consent
* Poor ear (ear to be implanted):

  * Pure-tone average (PTA) at .5, 1 and 2 kilohertz (kHz) > 70 dB HL (hereafter referred to as severe to profound hearing loss - SPHL)
  * Aided word recognition score (CNC Word Test) at 60 dB SPL ≤ 30%
  * Duration of SPHL ≥ 6 months
  * Onset of hearing loss ≥ 6 years of age
* Better ear:

  * PTA at .5, 1, 2, 4 kHz of 40 to 70 dB HL
  * Currently using a HA
  * Aided word recognition score (CNC Word Test) at 60 dB SPL > 40%
  * Stable hearing for the previous 1-year period. "Stable" is defined as thresholds that have not changed by more than 10 dB at 2 or more octave interval audiometric frequencies

Exclusion Criteria:

* Medical condition that contraindicates surgery
* Actively using an implantable device in the ear to be implanted
* Known cochlear malformation or obstruction that would preclude full insertion of the electrode array in the ear to be implanted
* Hearing loss of neural or central origin
* Unrealistic expectations related to the benefits and limitations of cochlear implantation
* Unwillingness or inability to comply with all investigational requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-07-28 (Actual); Primary Completion 2020-11-17 (Actual); Study Completion 2021-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill B Firszt, PhD, Principal Investigator — Washington University School of Medicine
Locations (4):
- United States (4):
  - House Clinic, Los Angeles, California
  - Saint Luke's Midwest Ear Institute, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - New York University School of Medicine, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sampathkumar R, Kaehne A, Kumar N, Kameswaran M, Irving R. Systematic review of cochlear implantation in adults with asymmetrical hearing loss. Cochlear Implants Int. 2021 Nov;22(6):311-329. doi: 10.1080/14670100.2021.1936363. Epub 2021 Jun 14. PMID 34126876

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from Summer 2017 through 2019.
Period: Overall Study
Arm/Group | Cochlear Implantation
Started | 40
Completed | 39
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cochlear Implantation
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.96 (10.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 33
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40
Length of Deafness - Poor Ear [Mean (Standard Deviation); unit: years] | 10.18 (12.06)

OUTCOME MEASURES:

1. Primary Outcome: Change in Poor Ear Alone CNC Monosyllabic Word Understanding in Quiet
Description: Group mean difference in CNC monosyllabic word understanding score in quiet with the CI alone at 6 months post-implant compared to pre-implant with a hearing aid. (CNC scored on a scale from 0% to 100%; Higher scores are better.)
Time Frame: Pre-implant and 6 months post-implant
Population: 36 participants had both pre-implant and 6-month post-implant CNC scores for the poor ear alone.
Measure: Mean (Standard Error); unit: percentage of words correct
Arm/Group | Cochlear Implantation
Number analyzed (Participants) | 36
percentage of words correct
  Pre-Implant Mean | 0.09 (0.016)
  6 Month Post-Implant Mean | 0.53 (0.422)
  Group mean difference | 0.44 (0.039)
Statistical Analysis 1: Comparison: Cochlear Implantation; Mean difference in percent correct for CNC words at 6 months post-implant and pre-implant is reported; Test type: Superiority; p < 0.001, t-test, 2 sided — The threshold for statistical significance was <=0.05; t(35) = 11.29

2. Primary Outcome: Change in Poor Ear Alone Soundfield Thresholds
Description: Group mean difference in soundfield thresholds (dB HL average across frequency range) with the CI alone at 6 months post-implant compared to pre-implant with a hearing aid. (Measurable decibels in hearing level (dB HL) generally range from -10 dB to 120 dB; Lower levels are better.)
Time Frame: Pre-implant and 6 months post-implant
Population: 36 participants had both pre-implant and 6-month post-implant Soundfield thresholds for the poor ear alone.
Measure: Mean (Standard Error); unit: Decibels
Arm/Group | Cochlear Implantation
Number analyzed (Participants) | 36
Decibels
  Pre-Implant Mean | 54.95 (1.72)
  6 Month Post-Implant Mean | 26.54 (1.03)
  Group mean difference | 28.41 (1.68)
Statistical Analysis 1: Comparison: Cochlear Implantation; Mean difference in Soundfield thresholds (averaged across the frequency range in dB HL) at 6 months post-implant and pre-implant is reported; Test type: Superiority; p < 0.001, t-test, 2 sided — The threshold for statistical significance was <=0.05; t(35) = 16.947

3. Secondary Outcome: Change in Sound Localization
Description: Sound localization in RMS error at 6-months post-implant in the CI+HA (CI at poor ear; HA at better ear) condition compared to the pre-implant best aided condition. (Root Mean Error Scores in degrees of error can range from 0 to approximately 80 degrees. Chance level performance is 64 degrees. Lower scores indicate better performance.)
Time Frame: Pre-implant and 6 months post-implant
Population: 36 participants had both pre-implant and 6-month localization scores in the bilateral/bimodal condition
Measure: Mean (Standard Error); unit: degrees RMS error
Arm/Group | Cochlear Implantation
Number analyzed (Participants) | 36
degrees RMS error
  Pre-Implant Mean | 45.05 (2.79)
  6 Month Post-Implant Mean | 39.07 (1.57)
  Group Mean Difference | 5.99 (2.80)
Statistical Analysis 1: Comparison: Cochlear Implantation; Mean difference in degrees RMS error at 6 months post-implant and pre-implant is reported; Test type: Superiority; p < 0.05, t-test, 2 sided — The threshold for statistical significance was <= 0.05; t(35) = 2.14

4. Secondary Outcome: Change in AzBio Sentences at 50 Decibels (dB) Sound Pressure Level (SPL)
Description: Understanding of sentences at a soft presentation level at 6-months post-implant in the CI+HA (CI at poor ear; HA at better ear) condition compared to the pre-implant best aided condition. (Percent correct ranging from 0 to 100%; Higher scores indicate better performance.)
Time Frame: Pre-implant and 6 months post-implant
Population: Both pre-implant and 6-month post-implant data were available for 36 participants.
Measure: Mean (Standard Error); unit: percentage of words correct
Arm/Group | Cochlear Implantation
Number analyzed (Participants) | 36
percentage of words correct
  Pre-Implant Mean | 66.81 (4.56)
  6-month Post-implant Mean | 83.06 (3.14)
  Group mean difference | 16.25 (4.04)
Statistical Analysis 1: Comparison: Cochlear Implantation; Mean difference in percentage of understanding (words correct) at 6 months post-implant and pre-implant is reported; Test type: Superiority; p < 0.001, t-test, 2 sided — The threshold for statistical significance was <= 0.05; t(35) = 4.02

5. Secondary Outcome: Change in AzBio Sentence Scores at 60 dB SPL and 4-talker Babble at +8 dB Signal-to-noise Ratio (SNR)
Description: Group mean difference in understanding of sentences in noise at 6-months post-implant in the CI+HA (CI at poor ear; HA at better ear) condition compared to the pre-implant best aided condition. (Percent correct scoring ranging from 0 - 100%; Higher scores indicate better performance.)
Time Frame: Pre-implant and 6 months post-implant
Population: 36 participants had both pre-implant and 6-mongh post-implant AzBio scores in noise.
Measure: Mean (Standard Error); unit: percentage of words correct
Arm/Group | Cochlear Implantation
Number analyzed (Participants) | 36
percentage of words correct
  Pre-Implant Mean | 64.39 (4.16)
  6-Month Post-Implant Mean | 71.42 (3.87)
  Group Mean Difference | 7.03 (2.72)
Statistical Analysis 1: Comparison: Cochlear Implantation; Mean difference in AzBio sentence scores in noise at 6 months post-implant and pre-implant is reported; Test type: Superiority; p < 0.05, t-test, 2 sided — The threshold for statistical significance was <= 0.05; t(35) = 2.58

6. Secondary Outcome: Change in Bamford-Kowal-Bench Speech-in-Noise (BKB-SIN) Sentence Understanding With Noise to the Better Ear
Description: Group mean difference in BKB-SIN scores in noise (dB SNR) 6-months post-implant in the CI+HA (CI at poor ear; HA at better ear) condition compared to the pre-implant best aided condition. Speech is from the front and noise to the better ear. (Scores are the signal to noise ration in decibels for approximately 50% understanding and can range from -7.5 dB to 23.5 dB; Lower scores indicate better performance.)
Time Frame: Pre-implant and 6 months post-implant
Population: 36 participants had BKB-SIN scores for noise to the better ear at both the pre-implant and 6-month test intervals
Measure: Mean (Standard Error); unit: dB Signal-to-Noise Ratio
Arm/Group | Cochlear Implantation
Number analyzed (Participants) | 36
dB Signal-to-Noise Ratio
  Pre-implant mean | 6.61 (0.83)
  6-month post-implant mean | 4.06 (0.83)
  Group mean difference | 2.56 (0.81)
Statistical Analysis 1: Comparison: Cochlear Implantation; Mean difference in dB SNR for BKB-SIN sentences with noise to the better ear at 6-months post-implant and pre-implant is reported; Test type: Superiority; p < 0.01, t-test, 2 sided — The threshold for statistical significance was <= 0.05; t(35) = 3.16

7. Secondary Outcome: Change in AzBio Sentence Scores at 60 dB SPL for the Poor Ear Alone
Description: Group mean difference in AzBio sentence scores in quiet for the poor ear alone with the CI at 6-months post-implant compared to pre-implant with a hearing aid. (Scores are percent of words correct and can range from 0 to 100%; higher scores indicate better performance.)
Time Frame: Pre-implant and 6 months post-implant
Population: 36 participants had poor ear alone AzBio sentence scores at both the pre-implant and 6-month test intervals.
Measure: Mean (Standard Error); unit: percentage of words correct
Arm/Group | Cochlear Implantation
Number analyzed (Participants) | 36
percentage of words correct
  Pre-implant mean | 13.97 (2.75)
  6-month post-implant mean | 64.86 (4.96)
  Group mean difference | 50.89 (4.89)
Statistical Analysis 1: Comparison: Cochlear Implantation; Mean difference in AzBio sentence scores at 60 dB SPL for the poor ear alone at 6 months post-implant and pre-implant is reported; Test type: Superiority; p < 0.001, t-test, 2 sided — The threshold for statistical significance was <= 0.05; t(35) = 10.42

8. Secondary Outcome: Change in Hearing Handicap Inventory (HHIE)
Description: Inventory completed by participant regarding emotional and social consequences of hearing loss. Group mean difference in the total HHIE ratings at 6-months post-implant compared to pre-implant. (Ratings can range from 0 to 100; Lower scores indicate less perceived hearing handicap - lower scores are better.)
Time Frame: Pre-implant and 6 months post-implant
Population: 39 participants had completed the HHIE at both the pre-implant and 6-month post-implant test intervals.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cochlear Implantation
Number analyzed (Participants) | 39
score on a scale
  Pre-implant mean | 0.67 (0.03)
  6-months post-implant mean | 0.46 (0.04)
  Group mean difference | 0.21 (0.03)
Statistical Analysis 1: Comparison: Cochlear Implantation; Mean difference in HHIE reported scores at 6-months post-implant and pre-implant is reported; Test type: Superiority; p < 0.001, t-test, 2 sided — The threshold for statistical significance was <= 0.05; t(38) = 7.15

9. Secondary Outcome: Change in Health Utility Index (HUI3) Ratings
Description: Questionnaire completed by participant regarding ability/disability across several health dimensions. Group mean difference in HUI3 ratings (total score) at 6 months post-implant compared to pre-implant. (Scores can range from 0.0 to 1.0; Higher scores indicate greater perceived health/ability.)
Time Frame: Pre-implant and 6 months post-implant
Population: 39 participants completed the HUI3 at both the pre-implant and 6-month post-implant test intervals.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cochlear Implantation
Number analyzed (Participants) | 39
score on a scale
  Pre-implant mean | 0.51 (0.04)
  6-month post-implant mean | 0.66 (0.03)
  Group mean difference | 0.15 (0.03)
Statistical Analysis 1: Comparison: Cochlear Implantation; Mean difference in HUI3 ratings at 6 months post-implant and pre-implant is reported; Test type: Superiority; p < 0.001, t-test, 2 sided — The threshold for statistical significance was <= 0.05; t(38) = 4.34

10. Secondary Outcome: Change in Speech, Spatial and Sound Qualities (SSQ) by 6-months Post-implant
Description: Questionnaire completed by participant regarding impact of hearing loss on various listening situations. Group mean difference in SSQ ratings at 6-months post-implant compared to pre-implant. (Ratings can range from 0 to 10; Higher scores indicate greater perceived abilities.)
Time Frame: Pre-implant and 6 months post-implant
Population: 39 participants had SSQ ratings at both the pre-implant and 6-month test intervals.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cochlear Implantation
Number analyzed (Participants) | 39
score on a scale
  Pre-implant mean | 3.42 (0.23)
  6-month post-implant mean | 5.46 (0.22)
  Group mean difference | 2.03 (0.26)
Statistical Analysis 1: Comparison: Cochlear Implantation; Mean difference in ratings for the SSQ total score at 6 months post-implant and pre-implant is reported; Test type: Superiority; p < 0.001, t-test, 2 sided — The threshold for statistical significance was <= 0.05; t(38) = 7.71

11. Secondary Outcome: Change in Speech, Spatial and Sound Qualities (SSQ) by 12-months Post-implant
Description: Questionnaire completed by participant regarding impact of hearing loss on various listening situations. Group mean difference in SSQ ratings at 12-months post-implant compared to pre-implant. (Ratings can range from 0 to 10; Higher scores indicate greater perceived abilities.)
Time Frame: Pre-implant and 12 months post-implant
Population: 39 participants had SSQ ratings for both the pre-implant and 12-month post-implant test intervals. (These were not the same 39 who had SSQ ratings at both the 6-month and pre-implant test intervals.)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cochlear Implantation
Number analyzed (Participants) | 39
score on a scale
  Pre-implant mean | 3.37 (0.23)
  12-month post-implant mean | 5.37 (0.25)
  Group mean difference | 2.00 (0.25)
Statistical Analysis 1: Comparison: Cochlear Implantation; Mean difference in SSQ ratings at 12 months post-implant and pre-implant is reported; Test type: Superiority; p < 0.001, t-test, 2 sided — The threshold for statistical significance was <= 0.05; t(38) = 7.90

12. Secondary Outcome: Change in Satisfaction With Amplification in Daily Use (SADL)
Description: Questionnaire completed by participant regarding satisfaction of HA use (pre-implant) and bimodal (HA+CI) device use at 6 months post-implant. (Ratings can range from 1 to 7; Higher scores indicate greater satisifaction.)
Time Frame: Pre-implant and 6 months post-implant
Population: 39 participants completed the HA version of the SADL pre-implant and also the bimodal version at 6 months post-implant (a modification of the original SADL).
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cochlear Implantation
Number analyzed (Participants) | 39
score on a scale
  Pre-implant mean | 4.88 (0.12)
  6-month post-implant mean | 5.36 (0.15)
  Group mean difference | 0.48 (0.20)
Statistical Analysis 1: Comparison: Cochlear Implantation; Mean difference in SADL scores at 6 months post-implant and pre-implant are reported; Test type: Superiority; p < 0.05, t-test, 2 sided — The threshold for statistical significance was <= 0.05; t(38) = 2.31

13. Secondary Outcome: Change in Scores on the Communication Profile for the Hearing Impaired (CPHI)
Description: The CPHI was completed by participant's spouse/significant other indicating their perception of how well the participant communicates in various situations. Group mean difference in CPHI ratings at 6 months post-implant compared to pre-implant. (Ratings can range from 1 to 5; Higher scores indicate better communication abilities as perceived by the spouse/significant other.)
Time Frame: Pre-implant and 6 months post-implant
Population: 26 participants had a spouse or significant other who completed the CPHI at both the pre-implant and 6-month post-implant test intervals.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cochlear Implantation
Number analyzed (Participants) | 26
score on a scale
  Pre-implant mean | 2.27 (0.10)
  6-month post-implant mean | 3.50 (0.15)
  Group mean difference | 1.22 (0.17)
Statistical Analysis 1: Comparison: Cochlear Implantation; Mean difference in the CPHI scores at 6 months post-implant and pre-implant are reported; Test type: Superiority; p < 0.001, t-test, 2 sided — The threshold for statistical significance was <= 0.05; t(25) = 7.27

14. Secondary Outcome: Change in Hearing Impaired Impact - Significant Other Profile (HII-SOP) by 6 Months Post-implant
Description: Questionnaire completed by participant's spouse/significant other indicating their perception of the impact of the participant's hearing loss on the spouse/significant other. Group mean difference in HII-SOP scores at 6 months post-implant compared to pre-implant. (Scores can range from 0 - 100; Lower scores are better - less impact of the hearing loss on the spouse/significant other.)
Time Frame: Pre-implant and 6 months post-implant
Population: 26 participants had a spouse or significant other who completed the HII-SOP at both the pre-implant and 6 month post-implant test intervals.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cochlear Implantation
Number analyzed (Participants) | 26
score on a scale
  Pre-implant mean | 55.96 (4.71)
  6-month post-implant mean | 22.98 (4.63)
  Group mean difference | 32.98 (4.31)
Statistical Analysis 1: Comparison: Cochlear Implantation; Mean difference in HII-SOP scores at 6 months post-implant and pre-implant is reported; Test type: Superiority; p < 0.001, t-test, 2 sided — The threshold for statistical significance was <= 0.05; t(25) = 7.65

15. Secondary Outcome: Change in Bamford-Kowal-Bench Speech-in-Noise (BKB-SIN) Sentence Understanding With Noise to the Poor Ear
Description: Group mean difference in BKB-SIN scores in noise (dB SNR) 6-months post-implant in the CI+HA (CI at poor ear; HA at better ear) condition compared to the pre-implant best aided condition. Speech is from the front and noise to the poor ear. (Scores are the signal to noise ration in decibels for approximately 50% understanding and can range from -7.5 dB to 23.5 dB; Lower scores indicate better performance.)
Time Frame: Pre-implant and 6 months post-implant
Population: 36 participants had BKB-SIN scores for noise to the poor ear at both the pre-implant and 6-month test intervals
Measure: Mean (Standard Error); unit: dB Signal-to-Noise Ratio
Arm/Group | Cochlear Implantation
Number analyzed (Participants) | 36
dB Signal-to-Noise Ratio
  Pre-implant mean | 1.82 (0.72)
  6-month post-implant mean | 0.42 (0.78)
  Group mean difference | 1.40 (0.60)
Statistical Analysis 1: Comparison: Cochlear Implantation; Mean difference in the dB SNR scores for BKB-SIN sentences at 6 months post-implant minus pre-implant is reported; Test type: Superiority; p < 0.05, t-test, 2 sided — The threshold for statistical significance was <= 0.05; t(35) = 2.34

ADVERSE EVENTS:
Time Frame: Approximately 15 months, from enrollment until 12-month evaluation.
Arm/Group | Cochlear Implantation
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 8/40
Other Adverse Events (participants affected / at risk) | 11/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cochlear Implantation (N=40)
Stroke (Vascular disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1) — at surgical site
Coronary angioplasty and stint (Vascular disorders) | 1 (1)
Gall bladder removal (Gastrointestinal disorders) | 1 (1)
Nausea (General disorders) | 1 (1) — Result of anesthesia
Kidney stone removal (Renal and urinary disorders) | 1 (1)
Tear of medial meniscus (Musculoskeletal and connective tissue disorders) | 1 (1)
Heart bypass surgery (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cochlear Implantation (N=40)
Dizziness (Ear and labyrinth disorders) | 7 (7) — onset or worsening
Tinnitus (Ear and labyrinth disorders) | 2 (2) — onset or worsening
Swelling (Ear and labyrinth disorders) | 2 (2) — Swelling over the cochlear implant receiver/stimulator

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-27): https://cdn.clinicaltrials.gov/large-docs/20/NCT03052920/Prot_SAP_000.pdf